CLINICAL TRIAL: NCT03358121
Title: Asprosin Dynamics Relating to Serum Glucose Levels Under Controlled Alteration
Brief Title: Glucose-dependent Asprosin Dynamics
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Stefan Kopf MD, Head of the Clinical Study Center for Diabetes Research, Heidelberg University
Other Study IDs: S-550/2016
Record Dates: First submitted 2017-10-26; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biobank, including serum and EDTA plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetics without hypoglycemia awareness: Diabetic patients without impaired hypoglycemia awareness. No interventions were performed, the study is purely observational.
  Interventions: Diagnostic Test: Clamp study
- Diabetics with hypoglycemia awareness: Diabetic patients with impaired hypoglycemia awareness. No interventions were performed, the study is purely observational.
  Interventions: Diagnostic Test: Clamp study

INTERVENTIONS:
Diagnostic Test: Clamp study — Clamp study to achieve high, normal, and lower glucose levels to study the dynamics of Asprosin.

SUMMARY:
The study entitled " Asprosin Dynamics relating to serum Glucose levels under controlled alterations" investigates the dynamics of Asprosin in relation to glucose levels under controlled conditions in diabetic patients.

DETAILED DESCRIPTION:
The Pilot study entitled Asprosin Dynamics relating to serum Glucose levels under controlled alterations is designed to date the asprosin kinetics at various metabolic states relating to serum glucose and the correlation between asprosin and the known glucose regulating hormones. Asprosin is the C-terminal cleavage product of profibrilln. This new hormone is encoded by FBN1 Gen (Amino acid residues 2732 to 2871, molecular weight 30 kDa), which also encodes fibrillin. The hormone was initially discovered during the analysis of the genome of patients with the extremely rare Wiedemann Rautenstrauch syndrome. According to the data so far, asprosin is a fast induced protein hormone that acts on the liver through cell membrane receptors, where it activates the G protein cAMP PKA pathway, leading to a rapid release of glucose into the circulation and to compensatory insulin production. The above seems to match the constellation found in overweight type 2 diabetes patients or patients with metabolic syndrome (insulin resistance). Diabetic mice were able to normalize their glucose and insulin levels by asprosin-binding antibodies. According to a recent study, asprosin had no influence on the serum concentration of glucagon, epinephrine, norepinephrine and cortisol in mice. In humans it is known that asprosin increases during fasting.

The liver related glucose release into the blood circulation is crucial for the brain function and overall survival during fasting. In addition, a compensatory rise in asprosin is expected during a hypoglycemic episode. In this pilot study, the asprosin concentration is measured both in participants with type 1 Diabetes mellitus, with or without hypoglycemia unawareness during a hypoglycemic phase. These relevant measurements are compared in the two subgroups, consisting of 5 persons each. By correlating asprosin values with other regulating hormones, there is hope to better understand the pathomechanism of hypoglycemia unawareness. Recently discovered is that the recombinant asprosin administration in mice allows both the blood glucose and the insulin to rise. It is therefore very likely that further studying of asprosin could provide new insights into the (patho) physiology of the intermediary metabolism disorder.

According to the above, the following hypotheses arise:

Asprosin dynamics relating to serum Glucose levels under controlled alteration:

Asprosin, as fast induced protein hormone, increases serum levels in type 1 diabetics with or without diabetes late complications during a hypoglycemic phase. Asprosin increases serum levels more significantly in diabetics without hypoglycemia unawareness compared to diabetics with hypoglycemia unawareness. There is probably no correlation between asprosin and the previous known regulating hormones. In order to investigate these hypotheses, study participants will be initially profoundly examined in our Clinical Study Center regarding both their glycemic metabolical responses and the clinical findings relating to their possible micro- and macrovascular complications. In addition to this quality of life, well being, depression and neuropathic pain is going to be taken into account. This is to be the first study of its kind, in which plasma levels of asprosin is determined and Type 1 diabetics with and without hypoglycemia unawareness are thoroughly examined in order to identify possible differences and similarities for the better determination of the new hormone utilizing the framework of hyperinsulinemic Clamp Tests. The intention behind is to better understand the (patho) physiology of the hypoglycaemia unawareness, as well as to better characterize the physiological properties of asprosin

ELIGIBILITY:
Inclusion criteria for participants without hypoglycemia unawareness

* Age between 18 and 75 years
* BMI between 20 und 35 kg per m2
* Persons with manifest diabetes mellitus type 1 and diagnosis according to according to DDG guidelines 2011 oGTT, HbA1c more than 6.5 percent in the absence of adulteration of the HbA1c, over 200 mg per dl in the 2 hour value of the oGTT, fasting glucose more than 126 mg per dl, spontaneous glucose more than 200 mg per dl at least twice.

Inclusion criteria for participants without hypoglycemia unawareness

* Persons who are not aware of hypoglycemia symptoms at glucose levels above 50 mg per dl
* Age between 18 and 75 years
* BMI between 20 und 35 kg per m2
* Persons with manifest diabetes mellitus type 1 and diagnosis according to DDG guidelines 2011 oGTT, HbA1c more than 6.5 percent in the absence of adulteration of the HbA1c, over 200 mg per dl in the 2 hour value of the oGTT, fasting glucose more than 126 mg per dl, spontaneous glucose more than 200 mg per dl at least twice.

General exclusion criteria Secondary types of diabetes (ADA criteria type 3 B to H)

* Current pregnancy
* Acute infections or fever Immune-suppressant therapy
* Severe psychiatric diseases requiring treatment (for example personality disorders, schizophrenia, depression)
* Known alcohol or drug dependency
* Severe heart, kidney, or liver insufficiency NYHA stadium IV
* Non-diabetic liver disease (for example PBC, PSC, Wilson's disease, hemochromatosis, autoimmune hepatitis)
* severe peripheral artery disease (stadium IV)
* non-diabetic glomerulopathy
* Cancer or other malignant diseases within the last 5 years
* Infectious diseases like hepatitis B, C, E, or HIV
* Other severe autoimmune diseases
* Current participation in an interventional study
* Anemia or disorders of bone marrow Exclusion criteria for clamp study
* Past history of deep vein thrombosis or pulmonary embolism
* Routine laboratory test results less than 80 percent below lower reference value: Ferritin, iron, leucocytes, haemoglobin, hematocrit, RBC, platelets, blood alcohol levels.

Exclusion criteria for bioimpedance

* measurement Pacemaker or ICD
* Exclusion criteria for lung function testing Ignoring or non-understanding of the instructions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 diabetic patients, five with and five without impairment in hypoglycemia awareness were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Asprosin dynamics | during clamp study, five hours
  Euglycemic hyperinsulinemic clamp It is a scientific test for the determination tissue sensitivity to insulin. The asprosin kinetic in various hyperglycemic and euglycemic phases as well as the correlation between asprosin levels to the other known regulating hormones will be investigated.
  An intravenous glucose tolerance test takes place in the morning and the serum glucose is controlled. Afterwards glucose 20 percent and insulin solution normal insulin is infused in order to set serum glucose manually at a target value of 90 mg per dl. The same test is performed with a glucose serum level of about 60 mg per dl, corresponding to physiological fasting serum glucose values. This is done in order to be able to assess asprosin kinetics even at lower serum glucose levels. At the end of this last hour, blood tests for the hormone measurement are performed. The duration of the examination is approximately 5 hours. Measurement of Asprosin is analyzed by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Stef Kopf, MD, Principal Investigator — Head of the Clinical Study Center for Diabetes Research
Locations (1):
- Medizinische Klinik, University Hospital, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27087445

DOCUMENTS (2):
  • Study Protocol (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT03358121/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT03358121/SAP_001.pdf